CLINICAL TRIAL: NCT05673161
Title: Retrospective Evaluation of the Effect of Iron (Fe) Infusion on Complications in Anemic Patients Undergoing Thoracotomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Assoc Prof Dr, Ankara University
Other Study IDs: 2022/613
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency Anemia Treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anemia, treatment: anemic patients who had iron therapy
  Interventions: Other: iron
- anemia, no treatment: anemic patients who had no therapy

INTERVENTIONS:
Other: iron — iron treatment
  Groups: anemia, treatment

SUMMARY:
In patients who underwent thoracotomy due to lung malignancy; It is desired to investigate whether there is a difference in terms of postoperative results between those with and without anemia, and those with iron deficiency anemia (IDA) who underwent intravenous iron replacement and those who did not, according to the hemoglobin value in their preoperative examinations.

ELIGIBILITY:
Inclusion Criteria:

* thoracotomy patients

Exclusion Criteria:

* emergency cases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergone thoracotomy
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
number of patients who had postoperatiive complication | 3 days
  postoperative complication
number of patients who received blood products | 3 days
  use of blood product

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After publishing the manuscript